CLINICAL TRIAL: NCT02904551
Title: Free Gingival Grafts for Implants Exhibiting Lack of Keratinized Gingiva: a Prospective Controlled Randomized Clinical Study
Brief Title: Gingival Augmentation Around Implants During Maintenance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Se-Lim Oh, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HR-00051371
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2024-12-11 (Actual); Status verified 2019-08

CONDITIONS: Failure of Dental Implant Due to Lack of Attached Gingiva
Keywords: prospective study; free gingival graft; keratinized gingiva; dental implant

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Free gingival grafts
  Interventions: Procedure: Free gingival graft
- Control (Active Comparator): Oral prophylaxis
  Interventions: Procedure: Oral prophylaxis

INTERVENTIONS:
Procedure: Free gingival graft — After infiltration anesthesia, a recipient bed was prepared with a horizontal split-thickness incision made with a 15 stainless steel blade at the mucogingival junction (MGJ) on the facial side of the selected implants. An intermediate thickness (0.75 mm) graft was taken from the palate. The graft was sutured with 6-0 polypropylene suture at the recipient site. Co-Pak® was applied on the recipient site. Analgesics (over-the-counter Tylenol or Ibuprofen) were prescribed for 5-7 days. PeridexTM (3M, St. Paul, MN) was prescribed for 7-10 days. No antibiotics were prescribed in relation to the surgery.
  Other Names: Experimental
  Arms: Experimental
Procedure: Oral prophylaxis — Oral prophylaxis is a regular dental cleaning. Titanium periodontal curette and superfloss were used on implant sites. Stainless steel periodontal curettes and a piezo scaler were used for natural teeth.
  Other Names: Control
  Arms: Control

SUMMARY:
This prospective controlled randomized blind clinical study investigated 44 implants displaying lack of KG in 29 subjects. Fourteen subjects received FGGs followed by oral prophylaxis. Fifteen subjects in the control group did not receive FGGs. The width of KG, gingival recession (GR), pocket depths (PD), plaque index (PI) and gingival index (GI) were assessed at baseline, 6, 12, and 18 months. Changes in crestal bone levels, from baseline, were assessed at 18 months.

DETAILED DESCRIPTION:
The purpose of this study was to evaluate clinical and radiographic outcomes following free gingival grafts (FGGs) around implants with limited keratinized gingiva (KG) compared to oral prophylaxis without gingival augmentation.

This prospective controlled randomized blind clinical study investigated 44 implants displaying lack of KG in 29 subjects. Fourteen subjects received FGGs followed by oral prophylaxis. Fifteen subjects in the control group did not receive FGGs. The width of KG, gingival recession (GR), pocket depths (PD), plaque index (PI) and gingival index (GI) were assessed at baseline, 6, 12, and 18 months.

There was a significant gain in KG with a reduction in GR in the FGG group compared to controls at 6, 12, and 18 months. The mean PI and GI were significantly lower for the FGG group at 12 and 18 months.

ELIGIBILITY:
Inclusion Criteria:

1. less than 2 mm KG present on the facial side of implant
2. implant restoration is single unsplinted unit, and has been in function for at least 6 months with an opposing dentition.

Exclusion Criteria:

1. uncontrolled hypertension
2. diabetes mellitus (DM),
3. subjects with a history of a long-term (>6 months) use of corticosteroid
4. subjects currently taking bisphosphonates, or with a history of taking bisphosphonates regardless of route of administration
5. subjects on medications that cause gingival hyperplasia
6. smokers
7. pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Changes in the width of Keratinized Gingiva from baseline to 6, 12, 18 months | 6, 12, 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Se-Lim Oh, DMD, MS, Principal Investigator — University of Maryland School of Dentistry
Locations (1):
- Advanced General Dentistry at UMB DS, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared. The results will be published.